CLINICAL TRIAL: NCT04496154
Title: The Inflammasome and Dysfunctional Adipose Tissue: Why Should apoB-lipoproteins be Targeted in Humans
Brief Title: Omega-3 to Reduce Diabetes Risk in Subjects With High Number of Particles That Carry "Bad Cholesterol" in the Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: May Faraj, PDt, PhD (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, May Faraj, PDt, PhD, Professor, Institut de Recherches Cliniques de Montreal
Organization: Institut de Recherches Cliniques de Montreal (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-14 and 2014-756; NUT273741 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Insulin Sensitivity/Resistance; Inflammatory Response; Fatty Acids, Omega-3
Keywords: HyperapoB; ApoB-lipoproteins; White adipose tissue; NLRP3 inflammasome; Fat metabolism; Insulin sensitivity and secretion; Systemic inflammation; Eicosapentaenoic acid (EPA); Docosahexaenoic acid (DHA)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omega-3 fatty acids (Experimental): 3 oral softgels (600 mg EPA and 300 mg DHA / softgel), Triple Strength Omega-3 from Webber Naturals
  Interventions: Dietary Supplement: Omega-3 fatty acids (2.7 g/d, EPA:DHA, 2:1)

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids (2.7 g/d, EPA:DHA, 2:1) — Triple Strength Omega-3 from Webber Naturals

SUMMARY:
In this project, investigators explored the role of the particles that carry "bad cholesterol" in the blood (termed LDL) that are known to promote heart disease, in the promotion of type 2 diabetes (T2D) in humans. In specific, they investigated how these particles may induce the activation of an immune pathway in human fat tissue leading to multiple anomalies that favors T2D. They also explored whether omega-3 fatty acids, which are the type of fat found in fish oils can counterbalance the negative effects of LDL in fat tissue, thus providing a natural way to help reduce the risk for T2D in subjects with elevated blood LDL.

To do so, 41 subjects who were free of disease or medication affecting metabolism were enrolled at the Montreal Clinical Research Institute between 2013 and 2019 and were placed on an intervention with omega-3 fatty acids supplementation for 12 weeks (2.7 g/day, Triple Strength Omega-3 from Webbers Naturals). Investigators examined the effects of LDL and omega-3 on risk factors for T2D before and after the intervention in the whole body and specifically in fat tissue biopsies taken from the hip region. Eighty percent of the subjects who were enrolled into the study completed the intervention.

DETAILED DESCRIPTION:
Diabetes-attributed deaths, mostly type 2 diabetes (T2D), total more than 40,000 per year, out of which 80% are secondary to cardiovascular disease and stroke. Research from the investigators' lab and others suggests that elevated atherogenic apoB-lipoproteins, mostly low-density lipoproteins (LDL) may not be a mere consequence of T2D but also a cause. They reported that high numbers of apoB-lipoproteins (apoB) induce subcutaneous white adipose tissue (WAT) dysfunction and predict several risk factors for T2D in humans. However, mechanisms underlying LDL-induced abnormalities and nutritional approaches to target them remain unexplored.

Strong evidence implicates a specific innate immunity system, the NLRP3 inflammasome/ interleukin 1 beta (IL-1β) pathway in WAT dysfunction and associated T2D risk factors in mice and humans (NLRP3 for Nucleotide-binding domain and Leucine-rich repeat Receptor, containing a Pyrin domain 3). Preliminary evidence from the investigator's lab and their collaborator (Dr Maya Saleh, at McGill University) indicated that native apoB-lipoproteins activate the NLRP3 inflammasome leading to IL-1β secretion in murine bone marrow derived macrophages. On the other hand, fish-oil derived omega-3 fatty acids, eicosapentaenoic and docosahexaenoic acids (EPA and DHA), were reported to inhibit the NLRP3 inflammasome/ IL-1β pathway in immune cells.

Thus, the central hypothesis of this trial was that apoB-lipoproteins act as metabolic danger-associated molecular patterns that activate the NLRP3 inflammasome in WAT leading to WAT dysfunction and associated risks for T2D in humans. This can be treated by EPA and DHA supplementation.

The specific hypotheses examined in 2 parts of this trial, at baseline and post-intervention, were:

Part A: At baseline (mechanisms):

Primary hypothesis:

1. Compared to subjects with low plasma apoB, subjects with high plasma apoB have higher WAT NLRP3 inflammasome activity indicated by higher WAT IL-1β secretion.

   Secondary hypotheses:
2. WAT IL-1β secretion is associated with risk factors for T2D (WAT dysfunction, systemic inflammation, postprandial hypertriglyceridemia, insulin resistance and hyperinsulinemia).
3. Ex vivo, subjects' native LDL prime and/or activate the NLRP3 inflammasome in subjects' own WAT.

Part B: Post-intervention (treatment of the baseline mechanisms):

Primary hypothesis:

1. Compared to subjects with low plasma apoB, twelve-week supplementation with EPA and DHA induces a greater reduction in WAT IL-1β secretion in subjects with high plasma apoB eliminating baseline group-differences.

   Secondary hypotheses:
2. Compared to subjects with low plasma apoB, twelve-week supplementation with EPA and DHA induces a greater reduction in risk factors for T2D in subjects with high plasma apoB.
3. Twelve-week supplementation with EPA and DHA reduces the baseline associations of WAT IL-1β secretion with risk factors for T2D
4. Ex vivo, EPA and DHA inhibit LDL-induced priming and/or activation of subjects' WAT NLRP3 inflammasome.

Forty-one subjects (34% men) were enrolled in the study, of whom 33 subjects completed the 12-week omega-3 intervention (drop out/exclusion rate = 20%). For statistical analysis, subjects were stratified into 2 groups based on baseline median plasma apoB per sex. The 2 groups with high plasma apoB and low plasma apoB were characterized and compared for the primary and secondary outcomes at baseline and following the omega-3 intervention.

ELIGIBILITY:
Inclusion Criteria:

Men and post-menopausal women:

* Having a body mass index (BMI) > 20 kg/m2
* Aged between 45 and 74 years
* Having confirmed menopausal status (FSH ≥ 30 U/l)
* Non-smoker
* Sedentary (less than 2 hours of structured physical exercise (ex: sports club) per week)
* Low alcohol consumption: less than 2 alcoholic drinks/day

Exclusion Criteria:

* Subjects with elevated risk of cardiovascular disease (≥ 20% of calculated Framingham Risk Score) who require immediate medical intervention by lipid-lowering agents OR who cannot be placed on a 4 weeks wash-out period from their lipid-lowering medication at screening (i.e. upon admission to IRCM clinic).
* Subjects with systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg
* Prior history of cardiovascular events (like stroke, transient ischemic attack, myocardial infarction, angina, heart failure...)
* Prior history of cancer within the last 3 years
* Thyroid disease - untreated
* Type 1 or 2 diabetes or fasting glucose > 7.0 mmol/L
* Claustrophobia
* Anemia - Hb < 120 g/L
* Creatinine > 100 μmol/L
* Hepatic dysfunction - AST/ALT > 3 times normal limit
* Blood coagulation problems (i.e. bleeding predisposition)
* Autoimmune diseases
* Chronic inflammatory diseases
* Concomitant medications

  * Hormone replacement therapy (except thyroid hormone at a stable dose)
  * Systemic corticosteroids
  * Anti-psychotic medications - psycho-active medication
  * Anticoagulant treatment (Aspirin, NSAIDs, warfarin, coumadin..)
  * Adrenergic agonist
  * Anti-hypertensive
  * Weight-loss
* Known substance abuse
* Allergy to seafood or fish
* Cancellation of the same scheduled testing visit, twice
* Lack of time to participate in the full length of the study (18 weeks)
* Have exceeded the annual total allowed radiation dose (like X-ray scans and/or tomography in the previous year or in the year to come) according to the physician's judgement.
* All other medical or psychological conditions deemed inappropriate according to the physician

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Fasting WAT IL-1β secretion | Baseline
  Accumulation of IL-1β in WAT medium ex vivo (by AlphaLISA)
Fasting WAT IL-1β secretion | At 12-weeks post-intervention
  Accumulation of IL-1β in WAT medium ex vivo (by AlphaLISA)

SECONDARY OUTCOMES:
WAT function and inflammation | Baseline
  Protein and gene expression of a panel of markers related to WAT function (e.g. ADIPOQ, PPARG, HMGCR, SREBP1C and 2) and inflammation (e.g. MCP1, ADGRE1, IL1B, NLRP3, IL10) by immunohistochemistry (relative to a total protein) and RT-qPCR (relative to HPRT).
WAT function and inflammation | Change at 12 weeks from baseline
  Protein and gene expression of a panel of markers related to WAT function (e.g. ADIPOQ, PPARG, HMGCR, SREBP1C and 2) and inflammation (e.g. MCP1, ADGRE1, IL1B, NLRP3, IL10) by immunohistochemistry (relative to a total protein) and RT-qPCR (relative to HPRT).
Postprandial fat metabolism | Baseline
  Area under the 6 hour time curve of plasma triglycerides after a high-fat meal (66% fat)
Postprandial fat metabolism | Change at 12 weeks from baseline
  Area under the 6 hour time curve of plasma triglycerides after a high-fat meal (66% fat)
Systemic inflammation | Baseline
  Fasting plasma inflammatory parameters including IL-1Ra
Systemic inflammation | Change at 12 weeks from baseline
  Fasting plasma inflammatory parameters including IL-1Ra
Insulin sensitivity and secretion | Baseline
  Glucose-induced insulin secretion and insulin sensitivity by Botnia clamps
Insulin sensitivity and secretion | Change at 12 weeks from baseline
  Glucose-induced insulin secretion and insulin sensitivity by Botnia clamps

OTHER OUTCOMES:
Plasma and red blood cells phospholipid fatty acid profile to assess compliance | Baseline
  by gas chromatography mass spectrometry
Plasma and red blood cells phospholipid fatty acid profile to assess compliance | Change at 12 weeks from baseline
  by gas chromatography mass spectrometry
Subject phenotyping | Baseline
  Fasting plasma metabolites (e.g. lipids, apoB) by COBAS INTEGRA, body composition (lean and fat mass in kg) by dual energy x-ray absorptiometry, total energy (kcal/day) and macronutrient intake (g/d) by 3-day dietary records and total energy (kcal/day) and macronutrient oxidation (g/d) by indirect calorimetry
Subject phenotyping | Change at 12 weeks from baseline
  Fasting plasma metabolites (e.g. lipids, apoB) by COBAS INTEGRA, body composition (lean and fat mass in kg) by dual energy x-ray absorptiometry, total energy (kcal/day) and macronutrient intake (g/d) by 3-day dietary records and total energy (kcal/day) and macronutrient oxidation (g/d) by indirect calorimetry
Post-hoc analysis of WAT receptors for apoB-lipoproteins and fatty acids | Baseline
  WAT surface-expression of LDLR and CD36 in WAT slides

CONTACTS AND LOCATIONS:
Overall Officials: May Faraj, PDt, PhD, Principal Investigator — Montreal Clinical Research Institute/ University of Montreal

IPD SHARING:
Plan to Share IPD: No
Biological samples (plasma and adipose tissue) can be made available for analysis by other investigators. However data statistical analysis incorporating complete IPD must be conducted by the research team of Dr May Faraj as per subject consent form.

REFERENCES:
- [Background] Lamantia V, Bissonnette S, Wassef H, Cyr Y, Baass A, Dufour R, Rabasa-Lhoret R, Faraj M. ApoB-lipoproteins and dysfunctional white adipose tissue: Relation to risk factors for type 2 diabetes in humans. J Clin Lipidol. 2017 Jan-Feb;11(1):34-45.e2. doi: 10.1016/j.jacl.2016.09.013. Epub 2016 Oct 3. PMID 28391908
- [Background] Bissonnette S, Saint-Pierre N, Lamantia V, Cyr Y, Wassef H, Faraj M. Plasma IL-1Ra: linking hyperapoB to risk factors for type 2 diabetes independent of obesity in humans. Nutr Diabetes. 2015 Sep 28;5(9):e180. doi: 10.1038/nutd.2015.30. PMID 26417659
- [Background] Lamantia V, Bissonnette S, Provost V, Devaux M, Cyr Y, Daneault C, Rosiers CD, Faraj M. The Association of Polyunsaturated Fatty Acid delta-5-Desaturase Activity with Risk Factors for Type 2 Diabetes Is Dependent on Plasma ApoB-Lipoproteins in Overweight and Obese Adults. J Nutr. 2019 Jan 1;149(1):57-67. doi: 10.1093/jn/nxy238. PMID 30535058
- [Background] Skeldon AM, Faraj M, Saleh M. Caspases and inflammasomes in metabolic inflammation. Immunol Cell Biol. 2014 Apr;92(4):304-13. doi: 10.1038/icb.2014.5. Epub 2014 Feb 11. PMID 24518981
- [Background] Lamantia V, Sniderman A, Faraj M. Nutritional management of hyperapoB. Nutr Res Rev. 2016 Dec;29(2):202-233. doi: 10.1017/S0954422416000147. Epub 2016 Nov 8. PMID 27821191
- [Background] Faraj M. LDL, LDL receptors, and PCSK9 as modulators of the risk for type 2 diabetes: a focus on white adipose tissue. J Biomed Res. 2020 Mar 12;34(4):251-259. doi: 10.7555/JBR.34.20190124. PMID 32701068
- [Result] Bissonnette S, Lamantia V, Ouimet B, Cyr Y, Devaux M, Rabasa-Lhoret R, Chretien M, Saleh M, Faraj M. Native low-density lipoproteins are priming signals of the NLRP3 inflammasome/interleukin-1beta pathway in human adipose tissue and macrophages. Sci Rep. 2023 Nov 1;13(1):18848. doi: 10.1038/s41598-023-45870-1. PMID 37914804
- [Result] Lamantia V, Bissonnette S, Beaudry M, Cyr Y, Rosiers CD, Baass A, Faraj M. EPA and DHA inhibit LDL-induced upregulation of human adipose tissue NLRP3 inflammasome/IL-1beta pathway and its association with diabetes risk factors. Sci Rep. 2024 Nov 7;14(1):27146. doi: 10.1038/s41598-024-73672-6. PMID 39511203